CLINICAL TRIAL: NCT04992936
Title: Effect of an Alcohol-Free Extract From the Wine Industry on Blood Pressure in Individuals With High Blood Pressure and Grade 1 Hypertension. Randomized, Crossover, Controlled Double Blind Study
Brief Title: Effect of an Extract From the Wine Industry on Blood Pressure (HYPERGRAPES)
Acronym: HYPERGRAPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: University Rovira i Virgili (Other); Grandes Vinos y Viñedos S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HYPERGRAPES
Record Dates: First submitted 2021-07-24; First posted 2021-08-05 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases; Hypertension
Keywords: Blood pressure; wine; by-products
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extract from the wine industry (Experimental): Participants will consume the extract from the wine industry for 5 weeks.
  Interventions: Dietary Supplement: Extract from the wine industry
- Placebo (Placebo Comparator): Participants will consume maltodextrin for 5 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Extract from the wine industry — The product will be presented in powder format in a single container and with a measuring spoon of the daily dose.
  Arms: Extract from the wine industry
Dietary Supplement: Placebo — The product will be presented in powder format in a single container and with a measuring spoon of the daily dose.
  Arms: Placebo

SUMMARY:
By-products from the wine industry pose serious problems of management, both from an economic and environmental point of view. Although traditionally the use of by-products of the wine sector has been limited to the production of biogas and energy, or its use as animal feed or agricultural fertilizer, there is greater interest in the use of these by-products as a potential source of functional ingredients.

Cardiovascular diseases (CVD) are the main cause of mortality in Europe, with hypertension being one of the main CVD risk factors. It has been shown that lowering blood pressure through behavioral and pharmacological interventions significantly improves CVD. Currently, one of the most widely used pharmacological therapies to treat hypertension is based on the use of angiotensin converting enzyme (ACE) inhibitors such as Captopril or Enalapril. ACE plays a key role in arterial pressure regulation, catalyzing the production of angiotensin II, an octapeptide with potent vasoconstrictor activity. In addition, ACE catalyzes the inactivation of bradykinin, peptide with vasodilator activity. The evaluation of various potential by-products of the wine industry for the generation of functional ingredients showed that an extract from the wine industry presented beneficial effects on blood pressure in in vitro models as well as in vivo models using rats with hypertension.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the effect of daily intake of an extract from the wine industry on the change in systolic blood pressure values in individuals with high blood pressure and grade 1 hypertension.

Secondary objectives are to evaluate the effects of an extract from the wine industry on:

* The change in diastolic blood pressure values.
* The change in body weight, body mass index (BMI) and waist circumference.
* The change in the circulating values of total cholesterol, LDL-c, HDL-c, triglycerides and ApoB.
* The change in the atherogenic index of plasma, which combines triglycerides and HDL-c values and which is considered a good indirect indicator of LDL-c particle size and subclinical atherosclerosis.
* Glucose metabolism and insulin resistance.
* The change in the inflammation values analyzed by the marker high sensitivity C-reactive protein.

Study Design: Randomized, crossover, placebo-controlled and double-blind nutritional intervention trial.

The number of subjects in the study will be 40. After the pre-screening visit, the participants will be randomly divided into two groups of 20 participants, according to start the study by taking the extract from the wine industry or placebo for 5 weeks. At the end of the week 5 of the study, when the first treatment is finished, there will be a washing period for 3 weeks and then the treatment will be changed for another 5 weeks: a total of 14 weeks.

The containers of the two treatments, the extract from the wine industry and the placebo, will present the same shape and appearance. The two products will present similar organoleptic characteristics of taste and color.

Each volunteer will make 5 visits, according to the crossover study design:

* a pre-selection visit (to check inclusion / exclusion criteria) (V0; week1) and, in case of meeting the inclusion criteria,
* two study visits during the consumption of the first product (extract from the wine industry or placebo), which will take place on the first day of study (V1; week 2) and after 5 weeks of treatment (V2; week 7).
* two study visits during the consumption of the second product (extract from the wine industry or placebo), which will take place after the three week washout period (V3; week 10) and after 5 weeks of treatment (V4; week 15).

In all visits except the V0 visit, participants must present themselves in fasting conditions of 8 hours to obtain blood. In addition, on V2 visits and V4 the participants will be asked the presence / absence of adverse effects that could be associated with the consumption of the study products.

Main variable: Systolic blood pressure levels.

Secondary variables:

* Diastolic blood pressure levels.
* Body weight.
* Height.
* Body mass index (BMI) (Kg/m2).
* Waist circumference.
* Conicity index.
* Waist circumference/Height ratio.
* Parameters in serum:
* Glucose.
* Insulin.
* Homeostatic Model Assessment for insulin resistance index (HOMA-IR).
* Total cholesterol.
* High density lipoproteins cholesterol (HDL-c).
* Low density lipoproteins cholesterol (LDL-c).
* Triglycerides (TG).
* Atherogenic indices:
* Total cholesterol/HDL-c
* LDL-c/HDL-c
* Plasma atherogenic index, calculated as the logarithm of the TG/HDL-c ratio.
* Apolipoprotein (apo) B.
* C-reactive protein.
* Faecal intestinal microbiota composition.
* Physical activity record.
* Record of potential adverse events.
* Frequency of consumption of supplements to avoid in the study.
* Completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age.
* Systolic blood pressure between 130- 159 mm Hg.
* Not under pharmacological treatment or have completed pharmacological treatment at least one month before the start of the study with anti-hypertensive and/or with lipid-lowering drugs. 2. Sign the informed consent.

Exclusion Criteria:

* BMI ≥ 35 kg/m^2.
* Have a clinical history of chronic kidney disease, cardiovascular disease and/or cancer.
* Be a smoker or ex-smoker in the last 6 months before inclusion in the study.
* Present diabetes.
* Take supplements with polyphenol components or aimed to lipid or blood pressure control during their participation in the study.
* Take 2 or more Standard Beverage Units daily or 17 weekly for women, or take 4 or more Standard Beverage Units daily or 28 weekly for men.
* Present some chronic gastrointestinal disease.
* Present food intolerances and/or allergies related to the products of the study, such as hypersensitivity to maltodextrin and/or sulfites.
* Being pregnant or intending to become pregnant.
* Be in breastfeeding period.
* Participate in or have participated in a clinical trial with drugs or nutritional intervention study in the last 30 days prior to inclusion in the study.
* Being unable to follow the study guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Systolic blood pressure will be measured using an automatic sphygmomanometer.

SECONDARY OUTCOMES:
Change in diastolic blood pressure | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Diastolic blood pressure will be measured using an automatic sphygmomanometer.
Change in body weight | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Body weight measured by standardized method.
Height | At week 1.
  Height measured by standardized method.
Change in BMI | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Weight and height will be combined to report BMI in kg/m^2.
Changes in waist circumference | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Waist circumference using a measuring tape.
Changes in conicity index | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Weight, height and waist circumference will be combined to report Conicity index.
Changes in waist circumference to height ratio | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Waist circumference and height will be combined to report Waist circumference to Height ratio.
Changes in serum glucose levels | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Serum glucose levels will be measured by standardized ultraviolet-visible spectrophotometry methods.
Changes in serum insulin levels | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Serum insulin levels will be measured by standardized chemiluminescence methods.
Changes in Homeostatic Model Assessment from Insulin Resistance Index (HOMA-IR) | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  HOMA-IR will be calculated using serum glucose and insulin levels.
Changes in serum total cholesterol levels. | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Serum total cholesterol levels will be measured by standardized ultraviolet-visible spectrophotometry methods.
Changes in serum HDL-c levels. | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Serum HDL-c levels will be measured by standardized ultraviolet-visible spectrophotometry methods.
Changes in serum LDL-c levels. | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Serum LDL-c levels will be calculated using the Friedewald formula.
Changes in serum Triglycerides levels | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Serum triglycerides levels will be measured by standardized ultraviolet-visible spectrophotometry methods.
Changes in total cholesterol to HDL-c ratio | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Total cholesterol and HDL-c values will be combined to report Total cholesterol to HDL-c ratio.
Changes in LDL-c to HDL-c ratio | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  LDL-c and HDL-c values will be combined to report LDL-c to HDL-c ratio.
Changes in Plasma atherogenic index | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Plasma atherogenic index will be calculated as the logarithm of the TG to HDL-c ratio.
Changes in serum Apo B levels | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Serum Apo B levels will be measured by standardized turbidimetry methods.
Changes in serum C- Reactive protein levels | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Serum C-Reactive protein levels will be measured by standardized turbidimetry methods.
Changes in intestinal microbiota composition | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Metagenomic analysis in fecal samples. The bacteria DNA will be extracted and massive sequenced by the Ion Torrent platform.
Change in Physical activity | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Physical activity will be evaluated through the International Physical Activity. Questionnaire (IPAQ)-short for physical activity questionnaire. The questionnaire asks about three specific types of activity (walking, moderate-intensity activities and vigorous intensity activities) in the set domains leisure time, domestic and gardening (yard) activities, work-related and transport-related activities. Frequency and duration are collected separately for each specific type of activity.
Adverse events | Before (baseline) and after treatment period (5 weeks) for each of the two treatments (dry VLC and placebo).
  Possible adverse events derived from taking study's products will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Del Bas, PhD, Principal Investigator — UTNS (Eurecat-Reus)
Locations (1):
- Eurecat, Reus, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with the Universitat Rovira i Virgili for the intestinal microbiota composition analysis
Supporting Information: Analytic Code
Time Frame: The data will be shared once the intervention period with the study participants has finished and will be shared until the end of the study analysis.
Access Criteria: The data will be encoded and access to the data will be controlled to only authorized personnel.

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org